CLINICAL TRIAL: NCT02015533
Title: A Randomized, Double-Blind, Placebo-Controlled Study in Healthy Japanese Subjects to Assess the Safety, Pharmacokinetics and Immunogenicity of CR8020 Following Single Intravenous Administration
Brief Title: A Study to Assess the Safety, Pharmacokinetics and Immunogenicity of CR8020 in Japanese Healthy Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to an unexpected preliminary result obtained from the study with CR8020.
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR102898; CR8020FLZ1002 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2013-12-13; First posted 2013-12-19 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2016-11

CONDITIONS: Healthy
Keywords: Healthy; CR8020; Japanese; Safety; Pharmacokinetics; Immunogenicity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CR8020 (Experimental)
  Interventions: Drug: CR8020
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CR8020 — CR8020 50 mg/kg solution will be administered as a single 2-hour intravenous infusion.
  Arms: CR8020
Drug: Placebo — Placebo will be administered as a single 2-hour intravenous infusion.
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess the safety, pharmacokinetics (what the body does to the drug) and immunogenicity (ability of a particular substance to provoke an immune response in the human body) of CR8020 in japanese healthy participants

DETAILED DESCRIPTION:
This study is a randomized (study medication is assigned by chance), double-blind (neither physician nor participant knows the treatment that the participant receives), placebo-controlled (placebo comparator is compared with the study medication to evaluate safety profile of the study medication in clinical study), single-dose study in Japanese healthy adult male participants. The study will include screening phase (28 to 2 days prior to the study medication administration), treatment phase (Study medication will be administered on Day 1), and follow-up phase (up to 99 days). Twelve participants will be randomly assigned to CR8020 50 mg/kg or placebo groups in a 2:1 ratio and receive an assigned treatment on Day 1. Safety will be assessed by evaluating adverse events, clinical laboratory tests, 12-lead Electrocardiogram, vital signs, and physical examination. Total maximum duration of participation of an individual participant will be 127 days.

ELIGIBILITY:
Inclusion Criteria:

* Have signed an informed consent document
* Body mass index between 18 and 30 kg/m2, with body weight greater than or equal to 50 kg at screening
* Must agree to use an adequate contraception method (eg, vasectomy, double-barrier, partner using effective contraception) and to not donate sperm from the study drug administration until Day 99
* Blood pressure between 90 and 140 mmHg systolic, inclusive, and no higher than 90 mmHg diastolic at screening
* Non-smoker or participant who smokes no more than 10 cigarettes, or 2 cigars, or 2 pipes of tobacco per day for at least 6 months before the study drug administration

Exclusion Criteria:

* History of or current clinically significant medical illness determined by the investigators including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, and coagulation disorders
* Clinically significant abnormal values for hematology, clinical chemistry or urinalysis
* Clinically significant abnormal physical examination, vital signs or 12-lead electrocardiogram
* A diagnosis of influenza infection or any constellation of clinical symptoms consistent with influenza infection within 14 days before the study drug administration is scheduled
* Participants with a fever of over 37.5°C on Day -1 or at predose

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to 99 days

SECONDARY OUTCOMES:
Maximum observed serum CR8020 concentration | Day 1 (predose, 0.5, 2.25, 4, and 8 hours), Day 2, Day 3, Day 4, Day 8, Day 15, Day 29, Day 43, Day 57, Day 71, Day 99 or early withdrawal day
Time to reach the maximum observed serum CR8020 concentration | Day 1 (predose, 0.5, 2.25, 4, and 8 hours), Day 2, Day 3, Day 4, Day 8, Day 15, Day 29, Day 43, Day 57, Day 71, Day 99 or early withdrawal day
Area under the serum CR8020 concentration-time curve | Day 1 (predose, 0.5, 2.25, 4, and 8 hours), Day 2, Day 3, Day 4, Day 8, Day 15, Day 29, Day 43, Day 57, Day 71, Day 99 or early withdrawal day
Level of antibodies to CR8020 in serum samples | Day 1 (predose), Day 29, Day 57, Day 99 or early withdrawal day
  Level of antibodies to CR8020 in serum samples will evaluate immunogenicity.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Osaka, Japan